CLINICAL TRIAL: NCT04271423
Title: Alveolar Ridge Preservation Using a Flap Versus Flapless Technique Using a Demineralized Bone Matrix Allograft Plus Mineralized Particulate Allograft and a Calcium Sulfate Barrier
Brief Title: Ridge Preservation Comparing a Flap Versus Flapless Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 047.06
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The flap procedure will consist of a full-thickness papilla preservation flap performed on the buccal and a full thickness flap on the palatal.
  Interventions: Procedure: Ridge Preservation
- Test (Experimental): The test will be a flapless technique, no flap will be reflected.
  Interventions: Procedure: Ridge Preservation

INTERVENTIONS:
Procedure: Ridge Preservation — Ridge Preservation using demineralized bone matrix and mineralized particulate allograft and covered with calcium sulfate barrier.

SUMMARY:
To compare a flapless technique of alveolar ridge preservation to a flap technique to determine if preserving the periosteal blood supply would prevent loss of crestal ridge width and height.

DETAILED DESCRIPTION:
Twenty-four patients will randomly be assigned to receive ridge preservation using either flapless or flap technique. Twelve test patients will receive ridge preservation using a flapless approach and twelve control patients will receive ridge preservation using a flap technique. All sockets will be grafted with demineralized bone matrix and mineralized particulate allograft and covered with calcium sulfate barrier. Re-entry surgery will be performed at 4 months when a trephine core will be taken from the grafted site immediately prior to implant placement and submitted for histologic processing.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced with a dental implant where at least one adjacent tooth is present
2. Study subjects at least 18 years old
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee of Institutional Review Board.

Exclusion Criteria:

1. Patients with debilitating systemic disease, or a disease affects the periodontium
2. Have an allergy to any material or medication used in the study
3. Require prophylactic antibiotics
4. Previous head and neck radiation therapy
5. Chemotherapy in the previous 12 months
6. Patients taking long term Non-steroidal Anti-inflammatory Drugs or steroid therapy
7. Smoked more than one pack of cigarettes per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Crestal Horizontal Ridge Width | 4 months after surgery
  Changes in post-extraction to 4 month change in ridge measurements at the alveolar crest and 5 mm apical to crest. Measurements taken with a caliper.

SECONDARY OUTCOMES:
Percent osseous tissue | 4 months after surgery
  A trephine core will be harvested at 4 months. Following histologic processing the osseous core will be classified into percent vital bone, nonvital bone and trabecular space

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville

IPD SHARING:
Plan to Share IPD: No